CLINICAL TRIAL: NCT06282666
Title: Comparison of Continuous Lumbar Erector Spinae Plane Block to Continuous Epidural Analgesia in Patients Undergoing Hip Replacement Surgery
Brief Title: Lumbar ESPB in Hip Replacement Surgery
Acronym: ESPB_HIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Michał Borys, MD, PhD, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KE-0254/150/2019
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Coxarthrosis; Pain, Postoperative; Pain, Acute; Pain, Chronic; Postoperative Pain, Chronic; Analgesia; Quality of Life; Anesthesia; Spinal
Keywords: erector spinae plane block; epidural analgesia; quality of recovery; patient-controlled analgesia; Timed Up and Go test; visual analog scale; neuropathic pain symptom inventory; Lovett scale; spinal anesthesia
MeSH Terms: conditions — Osteoarthritis, Hip; Pain, Postoperative; Acute Pain; Chronic Pain; Agnosia | interventions — Anesthesia, Spinal; Analgesia, Epidural; Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis; Visual Analog Scale; Sitting Position; Walking

STUDY DESIGN:
Intervention Model Description: Two groups will be randomly allocated to Epidural and ESPB (1:1)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will not be aware of the type of continuous blockade. Care providers, including doctors and nurses, will not be aware of patient allocation.
  Physiotherapists assessing outcomes will not be aware of patient allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural (Experimental): Combined spinal and epidural anesthesia will be performed before the surgery in the patient's lateral position with the operated hip down. The Espocan set will be used (B.Braun). After identification of the epidural space on the level of L3/L4, 0.5% bupivacaine (Marcaine Heavy Spinal) with fentanyl (5 mcg/mL) will be injected through the 27 G pencil point spinal needle. Then, the epidural catheter will be placed and a test dose of 2% lidocaine (2 mL) will be administered. At the end of the surgery, the patient will receive 5 mL of a mixture containing 0.1% bupivacaine with fentanyl (2 mcg/mL). Moreover, we will administer 5 mg of oxycodone i.v.
  the mixture of bupivacaine and fentanyl will be administered in a constant flow of 5 mL/h for a day.
  Interventions: Procedure: Spinal anesthesia; Procedure: Epidural analgesia; Procedure: patient-controlled analgesia; Diagnostic Test: Timed Up and Go test; Diagnostic Test: neuropathic pain symptom inventory; Diagnostic Test: Lovett test; Diagnostic Test: Visual analog scale; Diagnostic Test: Quality of Recovery 40; Diagnostic Test: Ability to sit, stand upright, and walk
- ESPB (Experimental): Spinal anesthesia will be performed in the patient's lateral position with the operated hip down. 0.5% bupivacaine (Marcaine Heavy Spinal) with fentanyl (5 mcg/mL) will be used and a 25-27 G pencil point spinal needle.
  The lumbar ESPB will be performed under ultrasound control at the L3 level on the ipsilateral site of the surgery. After dissection with 0.9 NaCl, a catheter will be left in the ESP. Then, we will administer 0.25% bupivacaine with epinephrine (5mcg/mL), 0.4 mL per kg, up to 40 mL. Moreover, 5 mg of oxycodone i.v. will be administered A mixture of 0.1% bupivacaine with fentanyl (2 mcg/mL) will be given in a constant flow of 5 mL/h for a day.
  Interventions: Procedure: Spinal anesthesia; Procedure: lumbar erector spinae plane block; Procedure: patient-controlled analgesia; Diagnostic Test: Timed Up and Go test; Diagnostic Test: neuropathic pain symptom inventory; Diagnostic Test: Lovett test; Diagnostic Test: Visual analog scale; Diagnostic Test: Quality of Recovery 40; Diagnostic Test: Ability to sit, stand upright, and walk

INTERVENTIONS:
Procedure: Spinal anesthesia — Before the beginning of surgery, all patients will be anesthetized with 0.5 % hyperbaric bupivacaine (Marcaine Heavy), 1.5 - 2.5 mL solution. A pencil point spinal needle will be used.
  Other Names: Subarachnoid anesthesia
Procedure: lumbar erector spinae plane block — Investigators will perform the lumbar ESPB under ultrasound control at the L3 level on the ipsilateral site of the surgery. After dissection with 0.9 NaCl, we will leave a catheter in the ESP. Then, we used 0.25% bupivacaine with epinephrine (5mcg/mL), 0.4 mL per kg, up to 40 mL.
  Other Names: ESPB
  Arms: ESPB
Procedure: Epidural analgesia — After identifying the epidural space and spinal anesthesia (combined technique), a catheter will be placed in the epidural space. Investigators will give an epidural catheter a test dose of 2% lidocaine (2 mL). At the end of the surgery, the patient will receive 5 mL of a mixture containing 0.1% bupivacaine with fentanyl (2 mcg/mL).
  Arms: Epidural
Procedure: patient-controlled analgesia — Each participant will receive a pump with oxycodone (1mg/ml) using a patient-controlled analgesia (PCA) technique, a bolus of 1 mL, and a lockout of 5 minutes for the first postoperative day.
  Other Names: PCA
Diagnostic Test: Timed Up and Go test — Investigators will measure the time the patient took to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while rotating 180 degrees. We will assess the patient before the surgery and 24 and 48 hours after hip replacement.
  Other Names: TUG
Diagnostic Test: neuropathic pain symptom inventory — The Neuropathic Pain Symptom Inventory (0-100; 0 denotes no pain, 100 the most severe pain) will be evaluated before the surgery and three and six months following the procedure.
  Other Names: NPSI
Diagnostic Test: Lovett test — A physiotherapist will use the six-grade Lovett scale to measure muscle strength, in which 0 denotes no muscle contractility, and 5 denotes the complete range of motion against gravity, with full resistance. We will test this before the surgery, 24 and 48 hours after the operation.
Diagnostic Test: Visual analog scale — Investigators will measure pain intensity with VAS (0-10; 0 denotes no pain, 10 maximal pain) before and after the surgery. Pain will be evaluated at rest and upon the activity.
  Other Names: VAS
Diagnostic Test: Quality of Recovery 40 — Investigators will assess the quality of recovery with QoR-40 a day after the surgery, a month, and three months following the procedure. The minimal score is 40, and the maximal is 200. The higher the result, the better the quality of recovery is.
  Other Names: QoR-40
Diagnostic Test: Ability to sit, stand upright, and walk — A physiotherapist will evaluate the patient's ability to sit, stand upright, and walk at planned times.

SUMMARY:
In this study, continuous erector spinae plane block (ESPB) will be compared to continuous epidural analgesia in patients undergoing elective hip replacement surgery. Opioid consumption, pain severity, quadriceps femoris muscle strength, ability to walk, and quality of recovery will be evaluated. Moreover, chronic pain severity in months after the hospital discharge will be assessed.

DETAILED DESCRIPTION:
This is a prospective trial in patients undergoing elective hip replacement surgery.

Written informed consent will be obtained from each patient, and our study will be conducted following the tenets of the Declaration of Helsinki for medical research involving human subjects.

Before the surgery, preoperative pain severity, chronic pain severity, and ability to sit, stand, and walk will be assessed.

Each participant will be anesthetized with spinal technique and randomly allocated patients according to postoperative analgesia to the continuous epidural (Epidural) group and the continuous lumbar erector spinae plane block (ESPB) group. Both regional techniques will be continued during the first day. Investigators will measure postoperative oxycodone consumption with a patient-controlled analgesia (PCA) pump. At several points, the patients' pain at rest and during activity will be evaluated on the visual analog scale (VAS, 0-10), their quadriceps femoris muscle strength on the Lovett scale (0-5), and their ability to sit, stand upright, and walk on the Timed Up and Go test. Moreover, the patient's recovery will be assessed through the Quality of Recovery 40 (QoR-40) questionnaire on the first postoperative day.

After the patient's discharge, information regarding acute and chronic pain severity and quality of recovery will be collected during the phone interview.

ELIGIBILITY:
Inclusion Criteria:

* primary hip replacement surgery due to coxarthrosis
* anesthetized with spinal technique
* able to use PCA pump
* having access to phone

Exclusion Criteria:

* patients taking painkillers not related to coxarthrosis;
* having active cancer,
* dementia or challenging contact with the patient;
* suffering from depression or other psychiatric disorders that required antidepressant treatment;
* consuming alcohol or recreational drug addiction;
* contraindications to the regional block.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Opiod consumtion with PCA | From the admission to the postoperative care unit to the next postoperative day for 24 hours.
  Oxycodone consumtion used with a patient-controlled analgesia pump

SECONDARY OUTCOMES:
Pain at rest | 24 hours before the surgery, after the surgery immediately in the postoperative care unit, 4, 8, 24, and 48 hours following the operation
  Pain measured at rest on the VAS (0-10)
Pain upon activity | 24 hours before the surgery, after the surgery immediately in the postoperative care unit, 4, 8, 24, and 48 hours following the operation
  Pain measured upon activity on the VAS (0-10)
Lovett test | 24 hours before the surgery, 24 and 48 hours after the operation
  The quadriceps femori's muscle strength on the Lovett scale (0-5)
TUG | 24 hours before the surgery, 24 and 48 hours after the operation
  Timed Up and Go test in seconds
QoR-40 | It will be measured 24 hours, 30 days, and three months following the surgery.
  quality of recovery 40
NPSI | 24 hours before the surgery and 3 and 6 months following the operation
  The Neuropathic Pain Symptom Inventory will be measured personally and after the discharge with a phone interview.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Piwowarczyk, M.D., Ph.D., Study Chair — Medical University of Lublin
Locations (1):
- II Department of Anesthesia and Intensive Care, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanych A, Kutnik P, Pasiak P, Zakrzewska-Szalak A, Wichowska O, Jednakiewicz M, Nogalski A, Piwowarczyk P, Borys M. Continuous lumbar erector spinae plane block as an alternative to epidural analgesia in pain treatment in patients undergoing hip replacement surgery - a prospective pilot study. Anaesthesiol Intensive Ther. 2023;55(4):272-276. doi: 10.5114/ait.2023.132517. PMID 38084571